CLINICAL TRIAL: NCT04063033
Title: Randomized Bilnded Controlled Trial Comparing The Effect of IV Sodium Ferric Gluconate Complex (FERRLECIT R) on Outcome Patients Admitted Due To Acute Decompansated Heart Failure With Iron Deficiency
Brief Title: IV Iron in Acute Decompensated Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Erez Marcusohn MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0290-19 RMB
Record Dates: First submitted 2019-08-18; First posted 2019-08-20 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — ferric gluconate

STUDY DESIGN:
Intervention Model Description: Randomisation to two groups, One receiving IV Iron on top of standard therapy while admitted to the hospital and the other receiving only standard therapy for acute heart failure.
Who Masked: Outcomes Assessor
Masking Description: Two cardiologists will examine the participants after 12 and 24 weeks and evaluate functional status and volume status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IV Iron treatment (Experimental): Patients will be administered IV Iron for 3-5 days. 125 mg per day.
  Interventions: Drug: IV iron - Sodium Ferric Gluconate Complex
- No IV Iron treatment (No Intervention): Patients will receive standard treatment for heart failure without IV Iron.

INTERVENTIONS:
Drug: IV iron - Sodium Ferric Gluconate Complex — IV Iron will be administered 125 mg each day, to 3-5 days during hospitalisation.
  Other Names: IV Ferrlecit
  Arms: IV Iron treatment

SUMMARY:
The study aims Compare the effect of addition of IV FERRLECITR (ferric gluconate) to standard therapy to standard therapy alone (without any IV iron treatment) in patients admitted with acute decompensated heart failure.

DETAILED DESCRIPTION:
Heart Failure (HF) constitutes one of the biggest burdens on the public health system, with incidence of 20 per 1000 persons above the age of 65 and up to 80 per 1000 persons above 85 years of age. Acute decompensated heart failure (ADHF) is the most common cause of hospitalizations among patients above the age of 65. Even with the advances in the treatment and management of HF, the prognosis of these patients remains poor. HF results in impaired quality of life (QoL), repeated hospitalizations and poor life expectancy.

Iron deficiency (ID) is a common comorbidity in HF patients, and is associated with poor outcome, worsening of New York Heart Association (NYHA) Class, and re-hospitalizations. While the mechanisms and pathophysiology of ID in HF is not well understood, it is presumed to be a combination of impaired absorption, renal dysfunction, hemodilution and drugs that are used for the treatment of HF.

The advantages of (intra-venous) IV ferric carboxymaltose to patients with reduced ejection fraction (HFrEF) with stable chronic heart failure and functional ID has been shown to reduce the risk of hospitalizations up to 60%, improve symptoms, exercise tolerance, functional capacity and overall QoL . Accordingly, the latest 2016 ESC Guidelines recommended the treatment in patients with HfrEF with reduced ejection fraction (HFrEF) and ID (Class IIA,LOC A).

The two major, placebo-controlled studies, mentioned above (CONFIRM-AF and FAIR-AF) have demonstrated the positive outcomes after correction of ID in stable HF patients, with a well-tolerated IV substance. However, there is no data today concerning the role of IV iron repletion in patients with decompensated HF and preserved EF. Furthermore, previous studies excluded a substantial portion of the HFrEF population recently admitted with (acute decompensated heart failure) ADHF and diagnosed with ID.

The effect of treating iron deficiency on quality of life an functional status has already been studied and found useful with various types of intravenous iron in the chronic kidney disease and inflammatory bowel disease.

In this study we aim to examine the effect of IV iron (ferric gluconate) which is a more affordable IV Iron on patients admitted due to acute heart failure with minimal exclusion criterias.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted due to acute decompensated heart failure to internal medicine department H or cardiology department.

   * Must meet two of the following criteria :

     * NT pro BNP > 300 pg/ml (>800 pg/ml in the presence of Atrial Fibrillation).
     * Peripheral pitting edema,
     * Jugular Venous Distention,
     * pulmonary edema/congestion according to physical examination or Chest X-ray.
   * IV furosemide treatment on admission to ER or internal ward/cardiology department.
2. Hb level 8-14 mg/dl on admission.
3. Iron stores: Ferritin <100 or Ferritin 100-300 and Transferrin saturation < 20%.
4. No evidence of active bleeding.
5. Patient provided informed consent.

Exclusion Criteria:

1. Cardiogenic shock or any other condition requiring IV vasopressors.
2. Previous allergy or anaphylaxis due to IV Iron.
3. Active malignancy undergoing treatment.
4. Status post major surgery involving substantial blood loss in the past 3 months.
5. Indication for Blood transfusion.
6. Infection indicating IV antibiotics.
7. History of acquired iron overload; known haemochromatosis or first relatives with hemochromatosis; and allergic disorders (asthma, eczema, and anaphylactic reactions).
8. hemolytic anemia.
9. History of chronic liver disease and/or alanine transaminase (ALT) or aspartate transaminase (AST) >3 times the upper limit of the normal range; chronic lung disease; myelodysplastic disorder; and known HIV/AIDS disease.
10. Recipient of immunosuppressive therapy or renal dialysis. History of erythropoietin, IV iron therapy, and blood transfusion in previous 30 days.
11. Unstable angina pectoris, as judged by the investigator; severe uncorrected valvular disease or left ventricular outflow obstruction; obstructive cardiomyopathy; uncontrolled fast atrial fibrillation or flutter (heart rate >110 beats per minute [bpm]); uncontrolled symptomatic brady- or tachyarrhythmias.
12. Musculoskeletal limitation that, in the judgement of the investigator, would impair cardiopulmonary exercise testing.
13. Pregnant or breastfeeding.
14. Inability to comprehend study protocol.
15. Parallel participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 12 and 24 Weeks
  The functional capacity will be evaluated by the 6 minute walk test at baseline,12 weeks and 24 weeks follow up.

SECONDARY OUTCOMES:
Change in NYHA | 12 and 24 weeks
  Change in NYHA from baseline to 12 and 24 weeks
All cause mortality | 1 Year
  Incidence of all cause mortality up to 1 year followup
Hospitalizations due to heart failure. | 1 year
  Incidence of hospitalisations due to heart failure up to 1 year followup

CONTACTS AND LOCATIONS:
Overall Officials: Erez Marcusohn, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marcusohn E, Borreda I, Hellman Y, Habib M, Bahouth F, Epstein D, Zukermann R. IV Sodium Ferric Gluconate Complex in Patients With Iron Deficiency Hospitalized due to Acute Heart Failure-Investigator Initiated, Randomized Controlled Trial. J Cardiovasc Pharmacol. 2022 Aug 1;80(2):194-196. doi: 10.1097/FJC.0000000000001287. PMID 35503997